CLINICAL TRIAL: NCT03299608
Title: Exhaled Breath Analysis for Rapid Diagnosis in Opportunistic Respiratory Infections in Hematological Patients
Brief Title: Rapid Analysis of Infections by Spectrometry of Exhaled Breath
Acronym: RAISE
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S60785
Record Dates: First submitted 2017-09-15; First posted 2017-10-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Respiratory Tract Infections; Hematologic Diseases
MeSH Terms: conditions — Respiratory Tract Infections; Hematologic Diseases | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Breath analysis — Spectrometric analysis of exhaled breath as screening for opportunistic respiratory infections

SUMMARY:
To quantify the diagnostic, prognostic and therapeutic value of spectrometric analysis of exhaled breath from hematological patients with respiratory infection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18y at start of study
* One of the following diagnoses:

  * De novo, refractory or relapsed AML/MDS receiving intensive chemotherapy
  * De novo, refractory or relapsed ALL/T-lymphoblastic lymphoma receiving intensive chemotherapy
  * Aplastic anemia requiring ATG therapy
  * Any patient admitted for either autologous hematopoietic stem cell transplantation. Transplantation may not have been performed at time of enrolment.
  * Any patient admitted with allogeneic hematopoietic stem cell transplantation within the last year, or planned during this admission.
* Written informed consent obtained from the patient

Exclusion Criteria:

* Hematological disease beyond the specified inclusion criteria
* Signs of active respiratory infection
* If previously enrolled: incomplete clearance of all signs of respiratory infection (both clinically, microbiologically and radiologically).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at high risk for opportunistic respiratory infections due to acute myeloid or lymphatic leukemia (undergoing intensive treatment), patients who underwent allogeneic stem cell transplantation, and patients receiving autologous stem cell transplantation
Sampling Method: Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | Through study completion (i.e. 6 weeks after diagnosis)
  Accuracy (expressed as specificity/sensitivity/NPV/PPV) will be assessed as compared to the revised EORTC-MSG criteria, at moment of diagnosis by high-resolution CT and bronchoscopy

SECONDARY OUTCOMES:
Diagnostic accuracy at 2 weeks as compared to the revised EORTC-MSG response criteria using high-resolution CT | 2 weeks after diagnosis
Diagnostic accuracy at 2 weeks as compared to the revised EORTC-MSG response criteria using high-resolution CT | 6 weeks after diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No